CLINICAL TRIAL: NCT07202624
Title: Evaluating the Effectiveness of Intracuff Dexmedetomidine Versus Alkalinized Lidocaine in Preventing Postoperative Sore Throat Following Prolonged Prone Surgery
Brief Title: The Effectiveness of Intracuff Dexmedetomidine in Preventing Postoperative Sore Throat Following Prone Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince Sultan Military Medical City (Other)
Responsible Party: Principal Investigator, Mohamed Daabiss, CONSULTANT ANESTHESIA, Principal Investigator, Prince Sultan Military Medical City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-01-R079
Record Dates: First submitted 2025-08-05; First posted 2025-10-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sore Throat
Keywords: Postoperative Sore Throat; Prone Surgery; Dexmedetomidine
MeSH Terms: conditions — Pharyngitis | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A, ETT cuff will be filled with dexmedetomidine (n = 50) (Experimental): ETT cuff will be filled with 4 ml of dexmedetomidine 4 mcg/ml.
  Interventions: Drug: Dexmedetomidine (Precedex)
- Group B, ETT cuff will be filled with alkalinized lidocaine (n = 50) (Active Comparator): lidocaine 2%, 2 ml will be initially injected into the cuff, and then a supplementary volume of 2 ml of sodium bicarbonate (NaHCO3) 8.4% will be added
  Interventions: Drug: alkalinized lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine (Precedex) — The ETT cuff will be filled with 4 mL of dexmedetomidine 4 mcg/mL
  Other Names: Group D
  Arms: Group A, ETT cuff will be filled with dexmedetomidine (n = 50)
Drug: alkalinized lidocaine — lidocaine 2%, 2 ml will be initially injected into the cuff, and then a supplementary volume of 2 ml of sodium bicarbonate (NaHCO3) 8.4% will be added
  Other Names: Group AL
  Arms: Group B, ETT cuff will be filled with alkalinized lidocaine (n = 50)

SUMMARY:
Postoperative sore throat (POST) is a common consequence of tracheal intubation, affecting 30% to 65% of patients, while hoarseness occurs in approximately 16% to 55% of cases. POST is undesirable as it negatively impacts the surgical experience, patient satisfaction, and daily activities even after discharge. It can result from factors such as vocal cord damage, nerve compression, blood loss, and injury to mucosal cells due to airway secretions and prolonged anesthesia.

Recent studies have identified several contributors to POST, including the shape and size of the tracheal tube, cuff pressure, duration of tube placement, and the use of inhalation anesthesia. Changing a patient's position from supine to prone can affect the cuff pressure and displacement of the endotracheal tube (ETT), which may influence the incidence of POST, hoarseness, and cough. Improper positioning can also strain neck muscles, putting pressure on the vocal cords and leading to hoarseness.

To reduce POST incidence, selecting the appropriate tracheal tube size is crucial, with recommended sizes of 6.0 to 7.5 mm for females and 7.0 to 8.0 mm for males. Maintaining cuff pressure between 20-25 mmHg is associated with a lower incidence of POST, as excessive pressure can cause mucosal trauma. Additional strategies include using video laryngoscopy for intubation, administering topical non-steroidal anti-inflammatory drugs (NSAIDs), and using steroids during surgery.

Recent research is exploring the effectiveness of intracuff saline and lignocaine for preventing coughing and POST. Increasing the alkalinity of local anesthetics with sodium bicarbonate can enhance their efficacy, improving diffusion through the ETT cuff. Dexmedetomidine, a selective alpha-2 receptor agonist, has shown promise in reducing cough rates and postoperative pain. Notably, a single dose of gargled dexmedetomidine (0.5 µg/kg) has demonstrated effects comparable to intravenous administration, and intratracheal dexmedetomidine has proven more effective than lidocaine in reducing cough reflex and facilitating smooth extubation.

DETAILED DESCRIPTION:
One hundred patients aged between 18 and 75 years, American Society of Anesthesiologists (ASA) physical status I and II patients of either sex, undergoing lumbar spine surgery in the prone position under general anesthesia with endotracheal intubation, will be prospectively investigated. Patients with a history of recent respiratory tract infection, prior medication with analgesics or corticosteroids will be excluded. Other Exclusion criteria will include patients who have preoperative sore throat, hoarseness, and cough, have a nasogastric tube, patients with Mallampati class > 2, and who required more than one attempt for tracheal intubation, or patients had a duration of tracheal intubation of < 60 min or > 300 min, and patients not willing to provide their voluntary written informed consent.

Using a computer-generated random number table, the patients will be randomly allocated into Group A, where the ETT cuff will be filled with dexmedetomidine (n = 50), or Group B, where the ETT cuff will be filled with alkalinized lidocaine (n = 50). An anesthetic nurse, who will not be taking part in the postoperative patient interview and assessment, will prepare the study solution and ETT.

In group A, the ETT cuff will be filled with 4 mL of dexmedetomidine 4 mcg/ml. While in group B, lidocaine 2%, 2 ml will be initially injected into the cuff, and then a supplementary volume of 2 ml of sodium bicarbonate (NaHCO3) 8.4% will be added to obtain the minimal occlusive volume. Patients will be premedicated with IV glycopyrrolate 0.2 mg and IV midazolam 0.03 mg/kg. Non-invasive blood pressure, electrocardiography, pulse oximetry, and patient state index (PSI) using a sedation monitor (SedLine, Masimo Corp, Irvine, CA 92618) will be applied when the patients arrive in the operating room. Anesthesia will be induced with fentanyl 2 μg /kg, propofol 2 mg/kg, and cisatracurium 0.2 mg/kg. The investigators will ventilate all patients with 100% oxygen via a facial mask. The investigators will perform tracheal intubation after confirming adequate muscle relaxation (the absence of movement and jaw relaxation). Endotracheal intubation will be performed with tubes having an internal diameter of 8.0 or 7.5 mm for male patients, and 7.5 or 7.0 mm for female patients.

One experienced anesthesiologist, blinded to the experimental protocol, will perform endotracheal intubation and anaesthesia in all patients during the study. Another anesthesiologist, who was not blinded to the study protocol, although excluded from the data collection, carefully inflated the cuffs in all patients. The cuff pressure will be inflated at the minimal occlusive volume i.e., no air leak around the tube cuff when positive pressure was administered at 20 cm. of water.

Patient's position will be changed from supine to prone for surgery, and the patient's head will be positioned on the sponge face pillow without head rotation. After the position change from supine to prone, the investigator will re-adjust the cuff pressure. Anesthesia will be maintained with 1.5-2.5 vol% sevoflurane and 50% in air. The end-tidal CO2 will be kept between 35 and 40 mmHg. The depth of anesthesia will be monitored and kept between 25 and 50 (PSI Index). units. Oral airway devices will not be used intraoperatively. Once the surgery is completed and the patient is fully awake (with TOF greater than 0.7 and PSI greater than 80), they will be extubated, followed by gentle oropharyngeal suction.

The primary outcome will be the incidence and severity of POST, and hoarseness and cough will be assessed for the 1st, 6th, 12th, and 24th hours after extubation. The assessment will be done by the on-call anesthesiology resident who was blinded to the study group. The severity of POST, hoarseness, and cough will be graded using a 4-point scale (0: no, 1: minimal, 2: moderate, 3: severe). Any patient who develops a post-operative sore throat will be given dexamethasone 8 mg IV stat and advised to perform warm normal saline gargles.

Postoperative visual analog scale scores (0 = no pain to 10 = the most severe pain). Fentanyl will be used to alleviate pain of a severity ≥5 on VAS through a bolus of 0.5 µg/kg. Episodes of nausea will also be assessed at each time point. Cricoid compression, duration of tracheal intubation, duration of prone position, duration of anesthetic time, and incidence of cough during extubation will be recorded.

The secondary objective will focus on monitoring hemodynamic parameters such as blood pressure, heart rate, and oxygen saturation. Measurements will be taken at multiple time points, including 5 minutes before anesthesia, baseline reading before tracheal intubation, 5 minutes post-intubation, every 15 minutes during surgery, and at 2, 12, and 24 hours following the procedure.

The sample size was estimated from preliminary data obtained from 40 patients, and the assumption that a 20% reduction in the incidence of POST would be clinically relevant.

The Power analysis suggested that a minimum of 44 patients in each group would be needed for a β = 0.2, α = 0.05, (adjusted Bonferroni's p-value). To compensate for potential dropouts (drop Rate = 10%), 50 patients will be enrolled in each group.

Data were analyzed using SPSS version 16.0 (SPSS Inc, USA) and will be presented as mean and standard deviation (SD) or frequencies (%). A parametric test (independent sample t-test) will be used for determining any difference between the means of two groups for a particular variable. Repeated measures analysis of variance (ANOVA) will be used to determine any difference in the basic monitoring profile and amount of drug required at different time intervals of individuals in both groups. A p-value <0.05 will be considered as statistically significant, and a p-value <0.001 as highly significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 75 years
* American Society of Anesthesiologists (ASA) physical status I and II patients
* Either sex
* Undergoing lumbar spine surgery in prone position under general anesthesia with endotracheal intubation.

Exclusion Criteria:

* Patients with a history of recent respiratory tract infection
* Prior medication with analgesics or corticosteroids.
* Patients who have preoperative sore throat, hoarseness and cough, have a nasogastric tube,
* Patients with Mallampati class > 2 and who required more than one attempt for tracheal intubation or patients had a duration of tracheal intubation of < 60 min or > 300 min and
* Patients not willing to provide their voluntary written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
the incidence and severity of POST, hoarseness, cough | Day 1 postoperative
  The primary outcome will be the incidence and severity of POST, hoarseness, cough will be assessed for 1st, 6th, 12th and 24th hour after extubation. The assessment will be done by the on-call anesthesiology resident who was blinded of the study group. The severity of POST, hoarseness, and cough will be graded using a 4-point scale (0: no, 1: minimal, 2: moderate, 3: severe) (Table 1) (15). Any patient will develop post-operative sore throat will be given dexamethasone 8 mg IV stat and advised warm normal saline gargles.

SECONDARY OUTCOMES:
hemodynamic parameters | Day 1 postoperative
  The secondary objective will focus on monitoring hemodynamic parameters such as blood pressure, heart rate, and oxygen saturation. Measurements will be taken at multiple time points, including 5 minutes before anesthesia, baseline reading before tracheal intubation, 5 minutes post-intubation, every 15 minutes during surgery, and at 2, 12, and 24 hours following the procedure.

OTHER OUTCOMES:
Weight in Kilograms, Height in meters | Day 1 postoperative
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Muteb AlOtaibi, MD, Study Chair — Prince Sultan Military Medical City
Locations (1):
- Prince Sultan Military Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Background] Aqil M, Khan MU, Mansoor S, Mansoor S, Khokhar RS, Narejo AS. Incidence and severity of postoperative sore throat: a randomized comparison of Glidescope with Macintosh laryngoscope. BMC Anesthesiol. 2017 Sep 12;17(1):127. doi: 10.1186/s12871-017-0421-4. PMID 28899338

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT07202624/Prot_SAP_000.pdf